CLINICAL TRIAL: NCT05268523
Title: Interventions to Teach Self-management Skills for Persisting Symptoms of COVID-19: Minimizing Impact of Symptoms on Everyday Functioning and on Healthcare Usage/utilization
Brief Title: Self-Management Interventions for Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: University Health Network, Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Robin Green, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-5038
Record Dates: First submitted 2022-03-03; First posted 2022-03-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: COVID-19
Keywords: Long-term effects; Self-management; Group therapy; Telerehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Single-Centre, multi-arm, pragmatic RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Education and Strategies Intervention Group (Experimental): Participants will use a videoconferencing system to participate in the Education and Strategies Intervention composed of 1 session per week (1.5 hrs/session) over the course of 8 weeks.
  Interventions: Behavioral: Education and Strategies Intervention
- Mindfulness Skills Intervention Group (Active Comparator): Participants will use a videoconferencing system to participate in the Mindfulness Skills Intervention composed of 1 session per week (1.5 hrs/session) over the course of 8 weeks.
  Interventions: Behavioral: Mindfulness Skills Intervention
- No-Treatment Control Group (No Intervention): Participants adhere to the standard of care (no study treatment) for 8 weeks.

INTERVENTIONS:
Behavioral: Education and Strategies Intervention — Sessions will be led by registered therapists and clinicians in the fields of psychology, rheumatology, cardiology and neurology. The sessions will be comprised of educational presentations on the nature of persisting symptoms after COVID-19 and associated recommendations for self-management.
  Arms: Education and Strategies Intervention Group
Behavioral: Mindfulness Skills Intervention — The Mindfulness Skills Intervention is an 8-week program designed to provide an introduction to some basic mindfulness skills. Each session begins with a brief breath focus practice followed by discussion of the experience and sharing/discussion of the previous week including participants' experiences. Each session also includes some didactics, and a new, related mindfulness skill is introduced and practiced, followed by another discussion.
  Arms: Mindfulness Skills Intervention Group

SUMMARY:
The purpose of this study is to investigate and compare the feasibility and efficacy of two group-based interventions (education vs. mindfulness) to help self-manage Long-COVID symptoms.

DETAILED DESCRIPTION:
After a COVID-19 infection, more than 75% of patients report ongoing somatic, cognitive, and psychiatric symptoms. At this time, research is needed to help develop treatments that limit the impact of these symptoms on people who have had COVID-19. The present study investigates the feasibility and efficacy of two group-based interventions in a single-centre, 3-arm, pragmatic RCT comprising (i) an Education Intervention Group arm, (ii) a Mindfulness Skills Intervention Group arm, and (iii) a No-Treatment Control Group arm. Phase 1 is a pilot RCT and will employ a mixed methods design with qualitative post-treatment interviews in a subset of participants in the Education Intervention Group arm only. Phase 2 is a full-scale, quantitative-only RCT, with refinements and power analysis based on the results of Phase 1. Sessions of both groups are delivered by licensed therapists and clinicians. Sessions last 1.5 hours per week for 8 weeks, with 10-15 patients/group in an online format. The Education group participants will learn about the nature of Long-COVID symptoms and discuss strategies for self-care/self-management of symptoms in recovery. The Mindfulness Skills Intervention group participants will receive an introduction to some basic mindfulness skills and practice strategies such as Mindfulness of Breath, Body, Sounds, Thoughts, and Choiceless Awareness.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed Long-COVID plus PCR positivity with and without hospitalization
* 3-12 months post-diagnosis of COVID-19
* >2 self-reported persisting symptoms in >1 mood, cognitive and/or somatic symptom domain
* Age >18
* English speaking
* Private access to computer/internet

Exclusion Criteria:

* Acute ventilator support
* Diagnosed dementia
* Past/present history of psychotic illness or mania and, because of potential overlap in symptoms, diagnosis of chronic fatigue syndrome, fibromyalgia, chronic lyme disease or traumatic brain injury
* Long-COVID symptom severity (i.e., physical, cognitive, emotional symptoms) at a level that would significantly interfere with attendance/adherence to the intervention protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Brief-COPE | Baseline and 1-week post-intervention.
  The Brief-COPE (Coping Orientation to Problems Experienced Inventory) is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Total scores are presented for three overarching coping styles as average scores (sum of item scores divided by number of items), indicating the degree to which the respondent has been engaging in that coping style (scores ranging from 1-4, where the higher the score, the better the coping ability). Increase in score is the better outcome, indicating improved coping ability.
Change in LOT | Baseline and 1-week post-intervention.
  The Life Orientation Test (LOT) is a 10-item scale that assesses one's dispositional level of optimism, coping and resilience. Respondents use a 5-point rating scale (0 = strongly disagree; 4 = strongly agree) to show how much they agree with 10 statements about positive and negative expectations. All scores are summed to obtain a total score from 0-24 with higher ratings meaning more optimism. Increase in score is the better outcome.
Change in Kessler Psychological Distress Scale (K10) | Baseline and 1-week post-intervention.
  This is a 10-item questionnaire measuring level of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period. Participant answer experiencing each feeling from 'none of the time' (score=1) to 'all of the time' (score=5). Scores of the 10 items summed to produce a total score between 10 and 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress. Decrease in score is the better outcome.
Change in SSS-8 | Baseline and 1-week post-intervention.
  The Somatic Symptom Scale - 8 (SSS-8) is a brief, 8-item self-report questionnaire used to assess somatic symptom burden. Participants rate how often they experience somatic symptoms (e.g. back pain, dizziness, headaches) on a scale from 0 (Not at all to) to 4 (Very much). Scores are summed to obtain total score between 0 and 32, the higher the score, the higher the somatic symptom burden. Decrease in score is the better outcome.
Change in Perceived Medical Condition Self-Management Scale | Baseline and 1-week post-intervention.
  The Perceived Medical Condition Self-Management Scale (PMCSMS) evaluates self-measured ability to manage a chronic health condition (Long COVID). Participants answer the 8 questions using a scale from 1-5, with 1 signifying "strongly disagree" and 5 signifying "strongly agree". All scores are summed to obtain a total score from 8-401 with higher ratings meaning better management. Increase in score is the better outcome.
Change in the Depression, Anxiety and Stress Scale | Baseline and 1-week post-intervention.
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) measures the emotional states of depression, anxiety and stress. Participants rate 21 emotional states on a scale of 0-3 to indicate how much the statement applied to them over the past week, with 0=never, to 3=almost always. Scores are summed to obtain total scores for each Depression, Anxiety and Stress category ranging between 0 and 21, the higher the score, the more severe the symptoms. Decrease in score is the better outcome.
Change in Quality of Life Enjoyment and Satisfaction Questionnaire | Baseline and 1-week post-intervention.
  TheQuality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a 16 item self-administered questionnaire that captures life satisfaction over the past week. Each question is rated on a 5 point scale from 1 (Very Poor) to 5 (Very Good). Scores from the individual items are added together and reported as percentage maximum possible score. The higher the score, the better the life enjoyment and satisfaction. Increase in score is the better outcome.
Change in Adapted Illness Intrusiveness Rating | Baseline and 1-week post-intervention.
  The Adapted Illness Intrusiveness Rating (AIIR) measures intrusiveness of symptoms in daily life. 13 items ask about how much Long-COVID and/or its treatment interferes with daily life on a scale of 1=not at all, to 7=very much. Scores are summed for domains of Physical Well-Being and Diet, Work and Finances, Marital, Sexual, and Family Relations, Recreation and Social Relations Items, Other Aspects of Life. The higher the total scores, the more intrusive the illness. Decrease in score is the better outcome.
Change in self-reported physician visits | Baseline and 1-week post-intervention.
  Participants will report how many times they have visited a physician during the past month. Answers will range from 0 to 10 or more. Reduction in the number of physician visits is the desired outcome.
Change in Self-efficacy | Baseline and 1-week post-intervention.
  The Self-Efficacy (Ages 18+) - Item Bank/Fixed Form is part of the measures in NIH Toolbox that measures self-efficacy, or the capacity to manage functioning and have control over meaningful events. Participants rate how often they experience events on a scale of 1=never to 4=very often. Items are summed to obtain total score. The higher the number, the higher their self-efficacy. Increase in score is the better outcome

SECONDARY OUTCOMES:
Feasibility: session feedback questionnaire | At the end of each weekly session for a duration of 8 weeks.
  Designed by our team, this session feedback questionnaires includes 3 questions asking the participant how useful and applicable they found the content taught during intervention sessions. Participants answer on a likert scale ranging from 1="Not at all useful" to 5="Very useful". Higher score is desired.
Feasibility: Recruitment rate | Collected during recruitment
  Determined by dividing the number of patients consented by the number of eligible patients approached. Rate closer to 1 is desired.
Feasibility: Retention rate | Collected during recruitment and 1 week post-follow-up
  Determined by dividing the number of consented patients at baseline by the number of consented patients retained at follow-up. Factors influencing retention (e.g., medical status) will be reported as percentages. Rate closer to 1 is desired
Feasibility: Adherence rate | Collected during each of the 8 session (1 sessions/week, 8 weeks)
  Determined by calculating the percentage of patients adhering to at least 80% of the training protocol. Compliance rates to be computed for individual participants weekly, and for full cohort at end of study. Rate closer to 100% is desired. Factors influencing recruitment, retention and completion will be documented and reported as percentages
Feasibility: qualitative interview | 1 week post-intervention
  Following an interview guide, participants will be asked two broad open questions, then probed for additional details. Participants will be asked about pros and cons of intervention design, then probed for further details based on the Workgroup for Intervention Development and Evaluation Research (WIDER) recommendations regarding content, format, delivery, timing issues and personnel. They will also discuss the impact of the intervention on health and health-related actions, then be probed for how the intervention affected self-management of Long-COVID symptoms and health care visits. A qualitative thematic analysis will be applied and key themes will be reported on.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Green, PhD, Principal Investigator — KITE- Toronto Rehabilitation Institute, University Health Network
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Gorna R, MacDermott N, Rayner C, O'Hara M, Evans S, Agyen L, Nutland W, Rogers N, Hastie C. Long COVID guidelines need to reflect lived experience. Lancet. 2021 Feb 6;397(10273):455-457. doi: 10.1016/S0140-6736(20)32705-7. Epub 2020 Dec 23. No abstract available. PMID 33357467
- [Background] Mahase E. Covid-19: What do we know about "long covid"? BMJ. 2020 Jul 14;370:m2815. doi: 10.1136/bmj.m2815. No abstract available. PMID 32665317
- [Background] Sykes DL, Holdsworth L, Jawad N, Gunasekera P, Morice AH, Crooks MG. Post-COVID-19 Symptom Burden: What is Long-COVID and How Should We Manage It? Lung. 2021 Apr;199(2):113-119. doi: 10.1007/s00408-021-00423-z. Epub 2021 Feb 11. PMID 33569660
- [Background] Taquet M, Geddes JR, Husain M, Luciano S, Harrison PJ. 6-month neurological and psychiatric outcomes in 236 379 survivors of COVID-19: a retrospective cohort study using electronic health records. Lancet Psychiatry. 2021 May;8(5):416-427. doi: 10.1016/S2215-0366(21)00084-5. Epub 2021 Apr 6. PMID 33836148
- [Background] Bryson WJ. Long-term health-related quality of life concerns related to the COVID-19 pandemic: a call to action. Qual Life Res. 2021 Mar;30(3):643-645. doi: 10.1007/s11136-020-02677-1. Epub 2020 Oct 18. PMID 33073307
- [Derived] Rybkina J, Jacob N, Colella B, Gold D, Stewart DE, Ruttan LA, Meusel LC, McAndrews MP, Abbey S, Green R. Self-managing symptoms of Long COVID: an education and strategies research protocol. Front Public Health. 2024 Feb 7;12:1106578. doi: 10.3389/fpubh.2024.1106578. eCollection 2024. PMID 38384879